CLINICAL TRIAL: NCT02013531
Title: Protocol 331-13-002: An Exploratory, Multicenter, Open-label, Flexible-dose Trial of Brexpiprazole (OPC-34712) as an Adjunctive Treatment in Adults With Major Depressive Disorder and Anxiety Symptoms
Brief Title: Brexpiprazole (OPC-34712) as an Adjunctive Treatment in Adults With Major Depressive Disorder and Anxiety Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-13-002
Record Dates: First submitted 2013-12-06; First posted 2013-12-17 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-02

CONDITIONS: Major Depressive Disorder; Anxiety
Keywords: schizophrenia; Major depressive disorder; Anxiety Symptoms; Mental Disorders; Psychotic Disorders; emotional withdrawal; antipsychotic
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Schizophrenia; Mental Disorders; Psychotic Disorders | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brexpiprazole (Experimental): Up to 3 mg/day, once daily dose, tablets, orally
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Treatment (6 weeks) - Up to 3mg/day, once daily dose, tablets, orally

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of flexibly dosed adjunctive brexpiprazole treatment in subjects with major depressive disorder and anxiety symptoms, who are experiencing an inadequate selective serotonin reuptake inhibitor (SSRI)/serotonin norepinephrine reuptake inhibitor (SNRI) response.

ELIGIBILITY:
Main Inclusion Criteria:

* Have a diagnosis of a single or recurrent, nonpsychotic episode of MDD as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and confirmed by both the Mini International Neuropsychiatric Interview (M.I.N.I.) and an adequate clinical psychiatric evaluation.
* Have a treatment history of an inadequate ADT response to at least 1 ADT (but not > 3) for the current episode.
* Have received a single, trial-approved, SSRI or SNRI at an adequate dose for

  ≥ 6 weeks prior to screening.
* Are 18 to 65 years old at the time of consent (inclusive, and outpatients only).
* Have a Hamilton Depression Rating Scale (HAM-D)-17-item Total Score ≥ 18 at screening and baseline.
* Have a Hamilton Anxiety Rating Scale (HAM-A) Total Score ≥ 20 at screening and baseline.

Main Exclusion Criteria:

Subjects with any of the following current Axis I DSM-IV-TR diagnoses:

* delirium
* dementia
* amnestic
* other cognitive disorders
* schizophrenia
* schizoaffective disorder
* other psychotic disorders
* bipolar I disorder,
* bipolar II disorder
* bipolar disorder not otherwise specified (NOS)
* eating disorders
* anorexia nervosa
* bulimia
* obsessive compulsive disorder
* post-traumatic stress disorder

Subjects with any of the following current Axis II DSM-IV-TR diagnoses:

* borderline, antisocial
* paranoid
* schizoid
* schizotypal
* histrionic personality disorders
* mental retardation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd Japan (OPCJ)
Locations (21):
- United States (21):
  - Tuscon, Arizona
  - Garden Grove, California
  - Oceanside, California
  - Temecula, California
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Lafayette, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Haverhill, Massachusetts
  - Rochester Hills, Michigan
  - New York, New York
  - Staten Island, New York
  - Salem, Oregon
  - Allentown, Pennsylvania
  - Arlington, Texas
  - Austin, Texas
  - Woodstock, Vermont
  - Richmond, Virginia

REFERENCES:
- [Derived] Weiss C, Meehan SR, Brown TM, Gupta C, Morup MF, Thase ME, McIntyre RS, Ismail Z. Effects of adjunctive brexpiprazole on calmness and life engagement in major depressive disorder: post hoc analysis of patient-reported outcomes from clinical trial exit interviews. J Patient Rep Outcomes. 2021 Dec 11;5(1):128. doi: 10.1186/s41687-021-00380-4. PMID 34894307
- [Derived] Davis LL, Ota A, Perry P, Tsuneyoshi K, Weiller E, Baker RA. Adjunctive brexpiprazole in patients with major depressive disorder and anxiety symptoms: an exploratory study. Brain Behav. 2016 Jul 24;6(10):e00520. doi: 10.1002/brb3.520. eCollection 2016 Oct. PMID 27781135

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 37 participants. 18 trial sites were initiated in the United Sates, and 12 trial sites enrolled participants.
Pre-assignment Details: The trial consisted of a 2- to 21-day screening phase, a 6-week (42-day) treatment phase, and a 30-day (+ 2) follow-up phase.
Groups:
- Brexpiprazole: Participants were administered oral brexpiprazole tablets of 0.5 milligram per day (mg/day) with titration up to 3 mg/day once daily (QD) in addition to their constant-dose ADT (anti-depressant therapy) for 6 weeks.
Period: Overall Study
Arm/Group | Brexpiprazole
Started | 37
Completed | 32
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Met Withdrawal Criteria | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Brexpiprazole: Participants were administered oral brexpiprazole tablets of 0.5 mg/day with titration up to 3 mg/day QD in addition to their constant-dose ADT for 6 weeks.
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is utilized as the primary efficacy assessment of a participant's level of depression. The MADRS consists of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items. The possible Total scores are from 0 to 60, with higher values indicating worse outcome.
Time Frame: Baseline, Week 6
Population: Participants took at least 1 dose of brexpiprazole and who had a valid Baseline and Post-Baseline efficacy assessment. A mixed model repeated measures (MMRM) analysis was performed.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Units on a scale | -19.6 (1.5)
Statistical Analysis 1: Comparison: Brexpiprazole; The null hypothesis of zero in mean change from Baseline in the MADRS total score at Week 6 was tested at a significance level of 0.05. Because this was an exploratory trial, no methods to control type I error rate were performed; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM with model terms: Baseline, visit, and Baseline by visit interaction

2. Secondary Outcome: Mean Change in Clinical Global Impression-Severity (CGI-S) Total Score
Description: The severity of illness for each participant was rated using the CGI-S. To perform this assessment, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Week 6
Population: Participants took at least 1 dose of brexpiprazole and who had a valid baseline assessment and Post-Baseline efficacy assessment. A MMRM analysis was performed.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Units on a scale | -2.2 (0.2)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 6; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed model repeated measure (MMRM) with model terms: Baseline, visit, and Baseline by visit interaction

3. Secondary Outcome: Mean Clinical Global Impression-Improvement (CGI-I) Score at Week 6.
Description: The improvement of each participants condition was rated for each participant using the CGI-I. The study physician rated the participants total improvement whether or not it was due entirely to drug treatment. To perform this assessment, the study physician answered the following question: "Compared to his/her condition at baseline, how much has the participant changed?" Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The response at a given week was compared with the participants condition at Baseline prior to the first dose of study medication.
Time Frame: Baseline, Week 6
Population: Participants took at least 1 dose of brexpiprazole and who had a valid baseline assessment and Post-Baseline efficacy assessment. The LOCF data set included data recorded at a scheduled treatment phase visit or, if no observation is recorded at that visit, data carried forward from the previous scheduled treatment phase visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Units on a scale | 1.9 (1.1)

4. Secondary Outcome: Percentage of Participants With CGI-I Response Rate
Description: as for outcome 3
Time Frame: Week 1 to Week 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
percentage of participants
  Week 1 | 8.3
  Week 2 | 36.1
  Week 3 | 50.0
  Week 4 | 66.7
  Week 6 | 75.0

5. Secondary Outcome: Percentage of Participants With a MADRS Response
Description: MADRS response rate, where response is defined as ≥ 50% reduction in respective total scores from Baseline to Week 6. The MADRS consists of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items. The possible Total scores are from 0 to 60, higher values indicate worse outcome.
Time Frame: Week 6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Percentage of participants | 69.4

6. Secondary Outcome: Percentage of Participants With a MADRS Remission
Description: MADRS remission rate, where remission is defined as MADRS Total Score ≤ 10 and 50% reduction in MADRS Total Score from Baseline to Week 6. The MADRS consists of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items. The possible Total scores are from 0 to 60, higher values indicate worse outcome.
Time Frame: Week 6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Percentage of participants | 47.2

7. Secondary Outcome: Mean Change From Baseline in Hamilton Depression Rating Scale (HAM-D17) Total Score
Description: The HAM-D17 was utilized as an assessment of a participants level of depression and was administered utilizing the Structured Interview Guide for the Hamilton Depression Rating Scale (SIGH-D). Detailed instructions for administration of this structured interview were provided in the SIGH-D. The HAM-D17 was administered at the following visits: screening, Baseline, and Week 6/ Early termination (ET). HAM-D17 is a 17-item questionnaire with a total score of 0 to 52 with higher scores indicating more depressive symptoms.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Units on a scale | -15.85 (7.37)

8. Secondary Outcome: Mean Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score
Description: The HAM-A was utilized for the evaluation of anxiety symptoms and was administered using the Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A). Detailed instructions for administration of this structured interview were provided in the SIGH-A. The HAM-A was administered at the following visits: screening, Baseline, Weeks 1, 2, 3, 4, and 6/ET. HAM-A is a 14-item scale with each item is scored on a scale from 0 (not present) to 4 (very severe) with a total score of 0 to 56, with higher scores indicating severe anxiety symptoms.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Units on a scale | -17.80 (1.23)
Statistical Analysis 1: Comparison: Brexpiprazole; The null hypothesis of zero in Mean change from Baseline in HAM-A total score at Week 6 was tested at a significance level of 0.05. Because this was an exploratory trial, no methods to control type I error rate were performed; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed model repeated measure (MMRM) with model terms: Baseline, visit, and Baseline by visit interaction

9. Secondary Outcome: Mean Change From Baseline in Sheehan Disability Scale (SDS) Mean Score
Description: The SDS was a self-rated instrument used to measure the effect of the participant's symptoms on work/school, social life, and family/home responsibilities. The SDS was a visual analogue scale that used spatio-visual, numeric, and verbal descriptive anchors simultaneously to assess disability across the 3 domains. The number most representative of how much each area was disrupted by symptoms was marked along the line from 0 = not at all to 10 = extremely. Scores of 5 and above were associated with significant functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Units on a scale | -3.62 (2.60)

10. Secondary Outcome: Mean Change From Baseline in Massachusetts General Hospital-Cognitive and Physical Functioning Questionnaire (MGH-CPFQ) Total Score
Description: The MGH-CPFQ was a participant-rated scale designed to assess cognitive and executive dysfunction including symptoms of fatigue in mood and anxiety disorders. The MGH-CPFQ consisted of 7 items, each rated on a scale from 1 (greater than normal functioning) to 6 (poorer than normal functioning). The total score of the 7 items ranged from 7 to 42, with higher scores indicative of a worse outcome. The MGH-CPFQ was administered at the following visits: Baseline and Week 6/ET.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Units on a scale | -9.85 (8.79)

11. Secondary Outcome: Mean Change From Baseline in Kellner Symptom Questionnaire (KSQ)
Description: KSQ is a subject-rated scale designed to assess distress using symptoms of depression, anxiety, anger-hostility and somatization. The questionnaire contains 92 items of which 68 items indicate symptoms and 24 items are antonyms of some of the symptoms that indicate well-being. The maximum score for each symptom subscale is 17, the well-being subscales 6 and for the total scale scores 23. A higher score indicates more distress than a lower score. The total subscale scores will be unevaluable if less than 19 of the 23 items are recorded. If 19 to 22 of the 23 items are recorded, the total subscale score is the mean of the recorded items multiplied by 23 and then rounded to the first decimal place. The total score will be unevaluable if less than 76 of the 92 items are recorded. If 76 to 91 of the 92 items and no less than 19 of the 23 items of each subscale are recorded, the total score will be the mean of the recorded items multiplied by 92 and then rounded to the first decimal place.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Units on a scale | -29.43 (20.88)

12. Secondary Outcome: Mean Change From Baseline in Go/No-Go Task for P-inhibition Failures
Description: Executive function and working memory were assessed for the Go/No-go Task using computer-based and paper-pencil neuropsychological instruments. These instruments focused on measuring impulse inhibition. The instrument was administered at the following visits: Baseline and Week 6/ET.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: failures
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 35
failures
  P-inhibition failures (Go cues) | -0.0193 (0.2324)
  P-inhibition failures (No-Go cues) | -0.0103 (0.2337)

13. Secondary Outcome: Mean Change From Baseline in Go/No-Go Task for Mean Reaction Time
Description: as for outcome 12
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 35
milliseconds
  Mean reaction time (Go cues) | -0.26 (52.49)
  Mean reaction time (No-Go cues) | -4.26 (51.69)

14. Secondary Outcome: Mean Change From Baseline in Delay Discounting Task - Monetary Choice Questionnaire (MCQ) Score
Description: Delay discounting was a participant-completed task is an index of impulsive behavior. It measured the extent to which the value of a reward decreased as the delay to obtaining that reward increased. The propensity of participants to delay reward was assessed with an MCQ. Discounting rate is estimated using, k= (A/V)1/D, where k is the discounting rate parameter, V is the immediate reward, A is the higher delayed reward and D is the amount of days to the delayed reward. The MCQ consists of 27 choices between immediate and delayed rewards. The participant chooses repeatedly between 2 hypothetical sums of money: a smaller amount now or a larger amount in the future (for example, "would you prefer $27 today or $50 in 21 days?") The answers provide an estimate of the participant's discounting rate; higher discounting rates indicate greater impulsivity. A total score is not computed for all 27 questions.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 35
unitless | -0.008442 (0.060200)

15. Secondary Outcome: Mean Change From Baseline in Delay and Probability Discounting Task (DPDT) Scores
Description: The experiential discounting task (EDT) was a subject-completed computerized task designed to measure delay discounting, an index of impulsive behavior. It measured the extent to which the value of a reward decreased as the delay to obtaining that reward increased. The participant chose between different amounts of money available at different delays or with different chances (probability to get the money). At the end of the session, one of the choices was selected at random, and the participant received whatever they chose in response of that question (immediate, delayed, or probabilistic amount). Formula for h-value: value = A / (1 + hO) p is probability of reward and O is odds against. The value of h indicates how the value of a reward and the probability of its occurrence decreases. The data are computerized and reflect delay discounting and impulsivity (higher discounting and higher probability discounting shows greater impulsivity). A total score is not computed for this task.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 29
unitless
  Delay discounting task k value | -3.586888 (15.156644)
  Probability discouting task h value | 3.505900 (28.036537)

16. Secondary Outcome: Mean Change From Baseline to Week 6 in the Number of Impulsive Choices in the Delayed Reward Task (DRT)
Description: Delay discounting was a participant-completed task considered as an index of impulsive behavior. It measured the extent to which the value of a reward decreased as the delay to obtaining that reward increased. During a training session, a single button with letter A or B appeared on the screen. The participant had to wait until the letter began to flash, and press the button only once. An amount of money was added to a counter and another single button appeared. During the test session, both buttons with letters A and B appeared on the screen. The participant had to choose one of the letters that remained; the other disappeared. The participant had to wait until the letter began to flash and then press the button again. An amount of money was added to the counter, and both letters appeared again. The data are computerized and reflect delay discounting and impulsivity (higher discounting shows greater impulsivity). A total score was not calculated for this task.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number of Impulsive Choices
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 35
Number of Impulsive Choices | 4.6 (18.1)

17. Secondary Outcome: Mean Change From Baseline in Food Delay Discounting Task
Description: Delay discounting was a participant-completed task considered as an index of impulsive behavior. The participant chooses between a reward they could have today and another that they could get after a specified amount of time. The participant would not receive the rewards, but was asked to make decisions as though he or she were really going to receive them. AUC is defined as area under the concentration-time curve; AUC for food is presented below. The data are computerized and reflect delay discounting and impulsivity (higher discounting shows greater impulsivity). To calculate the AUC, the "X-axis" is "days", "Y-axis" is "Food value", the actual area underneath the curve was calculated by summing the results for each delay and present value pair: x2 -x1[(y1 + y2)/2], where x1 and x2 are successive delays and y1 and y2 are the present values associated with those delays. The AUC can range from 1 (no discounting) to 0 (maximum discounting).
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 35
unitless | 0.0371 (0.1819)

18. Secondary Outcome: Mean Change From Baseline in Money Delay Discounting Task
Description: Delay discounting was a participant-completed task considered as an index of impulsive behavior. The participant chose between a reward they could have today and another that they could get after a specified amount of time. The participant would not receive the rewards, but was asked to make decisions as though he or she were really going to receive them. AUC is defined as area under the concentration-time curve; AUC for money is presented below. The data are computerized and reflect delay discounting and impulsivity (higher discounting shows greater impulsivity). To calculate the AUC, the "X-axis" is "days", "Y-axis" is "Money value", the actual area underneath the curve was calculated by summing the results for each delay and present value pair: x2 -x1[(y1 + y2)/2], where x1 and x2 are successive delays and y1 and y2 are the present values associated with those delays. The AUC can range from 1 (no discounting) to 0 (maximum discounting).
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 35
unitless | 0.0707 (0.2284)

19. Secondary Outcome: Mean Change From Baseline in Barratt Impulsiveness Scale 11-item (BIS-11) Total Score
Description: The BIS-11 was a participant-rated scale designed to assess impulsive personality traits. The BIS-11 consisted of 30 items scored on a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/always). The scores provided information to assess 6 first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and 3 second-order factors (motor impulsiveness, non-planning impulsiveness, and attentional impulsiveness). The total score ranged from 30 to 120, with higher scores indicating impulsive personality traits. The BIS-11 was administered at the following visits: Baseline and Week 6/ET.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 36
Units on a scale | -7.67 (10.14)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent until the follow-up visit of 30 (+2 days).
Groups:
- Brexpiprazole: Participants were administered oral brexpiprazole tablets of 0.5 mg/day to 3 mg/day, QD for 6 weeks.
Arm/Group | Brexpiprazole
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 28/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=37)
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=37)
Diarrhoea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 2
Influenza (Infections and infestations) | 2
Increased appetite (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Akathisia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No